CLINICAL TRIAL: NCT07285980
Title: Comparison of Bier Block and a Lidocaine-Propofol Mixture for the Prevention of Propofol Injection Pain: A Randomized, Double-Blind Clinical Trial
Brief Title: Comparison of Bier Block and Lidocaine-Propofol Mixture for Prevention of Propofol Injection Pain
Acronym: BBLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asma Ladib (Other)
Responsible Party: Sponsor-Investigator, Asma Ladib, Assistant Professor of Anesthesiology and Critical Care, University of Monastir
Organization: University of Monastir (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBLP2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Propofol Injection Pain
Keywords: propofol; lidocaine; Bier block; Intravenous regional anesthesia; Anesthesia, intravenous; Pain, injection
MeSH Terms: conditions — Pain | interventions — Propofol; Lidocaine

STUDY DESIGN:
Intervention Model Description: Three-arm parallel, randomized, double-blind clinical trial comparing the preventive efficacy of Bier block and lidocaine-propofol mixture on propofol injection pain.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the participant and the investigator assessing pain were blinded to group allocation. The propofol syringes were prepared by an anesthesiologist not involved in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group - Propofol alone (Active Comparator): Patients in this control arm received intravenous propofol at a dose of 2 mg/kg without any lidocaine pretreatment. Pain during propofol injection was evaluated, and results were used as the reference comparator for the two active investigational interventions.
  Interventions: Drug: propofol
- Lidocaine-Propofol Mixture Group (Experimental): Patients in this experimental arm received a mixture prepared by adding 40 mg of lidocaine directly into the propofol syringe immediately before intravenous administration. The total dose of propofol administered was 2 mg/kg. This intervention was evaluated relative to the control arm for its ability to reduce injection-related discomfort.
  Interventions: Drug: Lidocaine - Propofol Mixture
- Bier Block Group - Intravenous Lidocaine under Venous Occlusion (Experimental): Patients in this experimental arm received 40 mg of intravenous lidocaine administered under venous occlusion using a Bier block technique for approximately 2 minutes. After release of the tourniquet, propofol was administered intravenously at a dose of 2 mg/kg. This intervention was evaluated for its ability to reduce discomfort associated with propofol injection.
  Interventions: Drug: Lidocaine - Bier Block

INTERVENTIONS:
Drug: propofol — Intravenous anesthetic used for induction of anesthesia at a dose of 2 mg/kg.
  Other Names: Diprivan
  Arms: Control Group - Propofol alone
Drug: Lidocaine - Propofol Mixture — 40 mg lidocaine mixed directly with propofol prior to intravenous injection to reduce injection pain.
  Other Names: Xylocaine-Propofol mixture
  Arms: Lidocaine-Propofol Mixture Group
Drug: Lidocaine - Bier Block — 40 mg lidocaine injected intravenously under venous occlusion for 2 minutes before propofol administration.
  Other Names: Intravenous regional anesthesia with lidocaine
  Arms: Bier Block Group - Intravenous Lidocaine under Venous Occlusion

SUMMARY:
The goal of this clinical trial was to evaluate methods to prevent pain on intravenous administration of propofol during induction of anesthesia. Propofol frequently causes a burning or painful sensation when injected into a peripheral vein.

This randomized study compared three approaches in adult patients scheduled for elective surgery: propofol alone (control), propofol with 40 mg lidocaine mixed directly, and a brief intravenous lidocaine under venous occlusion (Bier block) using 40 mg for 2 minutes before propofol.

The primary outcome was the incidence of pain on propofol injection measured with a 4-point verbal rating scale (0 = no pain to 3 = severe pain). Secondary outcomes included pain intensity, peri-induction hemodynamic parameters, and local injection-site adverse effects.

DETAILED DESCRIPTION:
Study Design and Setting This study was designed as a prospective, single-center, randomized, double-blind, parallel-group clinical trial conducted at the Maternity and Neonatology Center of Monastir (Tunisia). The trial was carried out between March 2025 and July 2025 in accordance with institutional standards for general anesthesia.

Study Procedures Upon arrival in the operating room, standard monitoring was applied, including non-invasive blood pressure, electrocardiography, and pulse oximetry. A peripheral intravenous catheter was inserted in a vein of the upper limb used for propofol administration. No analgesic or sedative premedication was administered prior to induction.

Patients were allocated to one of three study groups according to a predefined randomization sequence. All study drugs were administered through the same intravenous access under standardized conditions.

In the control group, propofol was administered intravenously without lidocaine pretreatment. In the lidocaine-propofol mixture group, lidocaine was added directly to the propofol syringe immediately before injection. In the Bier block group, lidocaine was administered intravenously under venous occlusion using a tourniquet applied proximally for a short, predefined duration, followed by release of the tourniquet and intravenous administration of propofol.

Randomization and Blinding Randomization was performed using a block randomization method. Study syringes were prepared by an anesthesiologist not involved in patient management or outcome assessment. Patients, anesthesia providers, investigators, and outcome assessors remained blinded to group allocation throughout the study.

Data Collection and Monitoring Pain during propofol injection was assessed immediately at the time of administration by an independent observer using a standardized verbal rating scale. Hemodynamic parameters were recorded at predefined time points during induction of anesthesia. Patients were monitored for local adverse effects at the injection site following propofol administration.

Ethical Considerations The study was conducted in accordance with the principles of the Declaration of Helsinki. Ethical approval was obtained prior to study initiation, and written informed consent was obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* American Society of Anesthesiologists (ASA) physical status I to III
* Scheduled for elective surgery under general anesthesia requiring intravenous induction with propofol

Exclusion Criteria:

* Patient refusal
* Known hypersensitivity to local anesthetics or propofol
* Pre-existing vascular disease
* Infection at the intended injection site
* Chronic use of analgesics or anxiolytics
* Inability to understand the pain assessment scale
* History of drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pain during propofol injection | Immediate (within 30 seconds after propofol injection)
  Proportion of patients with any pain (score ≥1 on 4-point verbal rating scale).

SECONDARY OUTCOMES:
Severity of pain during propofol injection | Immediate (during propofol injection)
  Pain intensity on a 4-point verbal rating scale (0-3).
Change in mean arterial pressure after propofol injection | 1 minute after propofol injection
  Difference in mean arterial pressure between baseline and 1 minute after propofol injection.
Change in heart rate after propofol injection | 1 minute after propofol injection
  Difference in heart rate between baseline and 1 minute after propofol injection.
Local adverse effects at the injection site | Within 10 minutes after propofol injection
  Presence of erythema, edema, or venous irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Ladib, MD, Principal Investigator — Maternity and Neonatology Center of Monastir, Dept of Anesthesiology and Critical Care B
Locations (1):
- Maternity and Neonatology Center of Monastir, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (de-identified) that underlie the results reported in this article will be made available upon reasonable request to the principal investigator (Dr Asma Ladib, asmaladib@yahoo.com) after publication, for researchers who provide a methodologically sound proposal. Data will be available in an anonymized format for academic and non-commercial use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication, for 5 years
Access Criteria: Researchers with sound proposals may request anonymized data from Dr Asma Ladib for academic, non-commercial use